CLINICAL TRIAL: NCT06405672
Title: Comparison of Using an Endotracheal Tube With Stylet Versus an Endotracheal Tube Alone in Morbidly Obese Patients
Brief Title: The Effect of Endotracheal Tube With Stylet in Morbidly Obese Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 1/17
Record Dates: First submitted 2024-04-30; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Intubation; Difficult or Failed; Obesity, Morbid
Keywords: different intubation techniques; endotracheal tube; obesity; stylet
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotracheal tube with stylet (Other): The obese patients who will be intubated with stylet in laparoscopic sleeve gastrectomy
  Interventions: Procedure: Endotracheal tube with stylet
- Endotracheal tube alone (Other): The obese patients who will be intubated without stylet in laparoscopic sleeve gastrectomy
  Interventions: Procedure: Endotracheal tube alone

INTERVENTIONS:
Procedure: Endotracheal tube with stylet — The obese patients who will be intubated with stylet in laparoscopic sleeve gastrectomy
  Arms: Endotracheal tube with stylet
Procedure: Endotracheal tube alone — The obese patients who will be intubated without stylet in laparoscopic sleeve gastrectomy
  Arms: Endotracheal tube alone

SUMMARY:
The investigators aimed to compare the effects of using enotracheal tube with stylet versus endotracheal tube alone in morbidly obese patients undergoing sleeve gastrectomy.

DETAILED DESCRIPTION:
Different intubation techniques have been used in morbidly obese patients undergoing general anesthesia. No study comparing the use of endotracheal tube with or without stylet was found in literature. Thus, the investigators aimed to compare the effects of using enotracheal tube with stylet versus endotracheal tube alone in morbidly obese patients undergoing sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

Body mass index over 30 ASA physical status I-III Undergoing laparoscopic sleeve gastrectomy -

Exclusion Criteria:

Body mass index under 30 ASA physical status IV Unable to cooperate Refused to give writtten informed consent-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Intubation time | through study completion, an average of 6 months
  from handling laryngoscope to first vision of end-tidal CO2 waveform

SECONDARY OUTCOMES:
Intubation success | through study completion, an average of 6 months
  success or failure of first intubation attempt
complications | through study completion, an average of 6 months
  Undesirable complications such as laryngospazm, hoarseness will be recorded at postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Kerem İnanoğlu, MD, Principal Investigator — Antalya TRH

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaszynski T, Pietrzyk M, Szewczyk T, Gaszynska E. A comparison of performance of endotracheal intubation using the Levitan FPS optical stylet or Lary-Flex videolaryngoscope in morbidly obese patients. ScientificWorldJournal. 2014;2014:207591. doi: 10.1155/2014/207591. Epub 2014 May 20. PMID 24967423
- [Background] Nicholson A, Smith AF, Lewis SR, Cook TM. Tracheal intubation with a flexible intubation scope versus other intubation techniques for obese patients requiring general anaesthesia. Cochrane Database Syst Rev. 2014 Jan 17;2014(1):CD010320. doi: 10.1002/14651858.CD010320.pub2. PMID 24443105